CLINICAL TRIAL: NCT03932318
Title: A Phase I/II Study of Venetoclax and Azacitidine and Lintuzumab-Ac225 in Patients With Refractory or Relapsed AML
Brief Title: Venetoclax, Azacitidine, and Lintuzumab-Ac225 in AML Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study postponed
Sponsor: Actinium Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIN-AC225-AML03
Record Dates: First submitted 2019-04-17; First posted 2019-04-30 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia; Relapsed Adult AML
Keywords: Lintuzumab-Ac225; Venetoclax; Azacitidine; Lintuzumab; Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I and Phase II (Experimental): Lintuzumab-Ac225 will be administered on Day 8 of each cycle for four cycles (unless in the 0.5 μCi/kg or 0.25 μCi/kg cohorts, where there is a potential for an additional four cycles, pending PI and Medical Monitor review).
  Venetoclax will be taken on Days 1-21 of each cycle for up to 12 cycles.
  Azacitidine will be administered on Days 1-7 of each cycle for up to 12 cycles.
  Each cycle is 28 days, with a potential to expand to 42 days to allow for full hematologic recovery.
  Interventions: Biological: Lintuzumab-Ac225; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Biological: Lintuzumab-Ac225 — In the Phase I, patients will be enrolled into the following dose escalation cohorts: 0.50 μCi/kg, 1.0 μCi/kg, and 1.5 μCi/kg. If the 0.50 μCi/kg dose is determined to exceed the MTD, a 0.25 μCi/kg dose will be explored.
  Other Names: Actimab
Drug: Venetoclax — 400 mg daily will be taken orally on Days 1-21 of a 28-day cycle. There will be a ramp up of venetoclax dosing in the first cycle, with 100 mg administered on Day 1, 200 mg on Day 2, and 400 mg on Day 3 and Day 4 and later. Patients on antifungal azoles should receive one-half these doses, up to a maximum of 200 mg of venetoclax.
  Other Names: Venclexta
Drug: Azacitidine — 75 mg/m2 will be administered on days 1-7 of a 28-day cycle.
  Other Names: Vidaza

SUMMARY:
The study is a multicenter, open label Phase I/II trial.

1. To determine the maximum tolerated dose (MTD) of lintuzumab-Ac225 when given in combination with venetoclax and azacitidine for patients with CD33 positive AML. (Phase I portion)
2. To assess the percentage of patients with CR, CRh, CRi, MLFS or Overall Response (CR + CRh + CRi + MLFS), up to 6 months after the start of treatment without receiving other AML therapies.. (Phase 2 portion)

DETAILED DESCRIPTION:
The study is a multicenter, open label Phase I and Phase II trial combining lintuzumab-Ac225 with venetoclax and azacitidine in patients who have relapsed or refractory AML.

The Phase I portion is a dose-finding study which will enroll at least three patients at each dose level. Patients in each dose level will be observed for a minimum of 4 weeks before dose escalation occurs. There is no dose escalation for any individual patient. Lintuzumab-Ac225 is administered on Day 8 of the first 4 treatment cycles.

The Phase II portion of the study will enroll patients at the MTD dose level of lintuzumab-Ac225 as determined in the Phase I portion of the study. The goal of the Phase II portion will be to further characterize the safety and efficacy of the MTD dose of lintuzumab-Ac225.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed acute myeloid leukemia
2. Refractory or relapsed AML which will include:

   1. Refractory disease will be defined as at least 1 prior treatment with no remission.
   2. Relapsed disease will be defined as 5% or more blasts in bone marrow seen after remission.
   3. Patients with AML arising from myelodysplastic syndromes (including CMML) or myeloproliferative neoplasms (secondary AML, ts-AML) are also eligible.
3. White blood cell (WBC) count < 10 x 109/L;

   a. Use of hydroxyurea, prior to Cycle 1 and during Cycles 1 and 2, is permitted to lower the WBC count in the peripheral blood.
4. Age > 18 years.
5. Estimated creatinine clearance ≥ 50 mL/min calculated by the Cockroft-Gault formula.
6. AST and ALT ≤ 3.0 x ULN (unless considered to be due to leukemic organ involvement).
7. Bilirubin ≤ 3.0 x ULN (unless considered to be due to leukemic organ involvement).
8. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.

Exclusion Criteria:

1. Have acute promyelocytic leukemia (APL).
2. Active CNS leukemia. Patients with symptoms of CNS involvement, particularly those with M4 or M5 subtypes, should undergo lumbar puncture prior to treatment on study to exclude CNS disease. Symptoms include cranial neuropathies, other neurologic deficits, and headache.
3. Have received prior radiation to maximally tolerated levels to any critical normal organ.
4. Participant has received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of study treatment.
5. Clinically significant cardiac disease.
6. Active, uncontrolled serious infection.
7. Have other non-myeloid malignancy within 2 years of entry (with exceptions).
8. Psychiatric disorder that would preclude study participation
9. Previous solid organ transplant (prior treatment with SCT is allowed but not if patient as GVHD or is still receiving immunosuppression/GVHD therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) of Lintuzumab-Ac225 | Cycle 1, up to 48 days
  To determine the maximum tolerated dose (MTD) of lintuzumab-Ac225 when given in combination with venetoclax and azacitidine for patients with CD33 positive AML
Phase II: Overall Response (CR + CRh + CRi + MLFS) | Up to 6 months
  To assess the percentage of patients achieving CR, CRh, CRi, morphologic leukemia-free state (MLFS), or Overall Response (CR + CRh + CRi + MLFS), up to 6 months after the start of treatment without receiving other AML therapies

SECONDARY OUTCOMES:
Phase I: Overall Response | Up to 6 months
  Number of patients who's overall response is CR or CRh or CRi or MLFS
Phase I: OS | Phase I: End of 6 months, 12 months, 24 months.
  Number of patients who died
Phase II: OS | Phase II: End of 6 months, 12 months, 24 months
  Number of patients who died
Phase I and II: DFS | Through study completion, up to 2 years
  Disease-free survival
Phase I and II: Evaluate incidence of AEs and SAEs | Through study completion, up to 2 years
  Rate of AEs and SAEs, including infusion-related reactions
Phase I and II: Lab abnormalities (other than hematologic indices) | Through study completion, up to 2 years
  Summary of rate of Grade 3/4 lab abnormalities
Phase I and II: Evaluate BH3 priming assay results | Completion of Cycle 1, estimated 1 month
  Summary of assay results
Phase I and II: MRD status | From date of first dose until the date of first documented response, first assessment at 6 months
  Number of patients who are MRD negative

CONTACTS AND LOCATIONS:
Overall Officials: Avinash Desai, MD, Study Chair — Actinium Pharmaceuticals, Inc.